CLINICAL TRIAL: NCT05091112
Title: Nerve Composition of Human Lumbar Dorsal Primary Rami and Its Medial Branch
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 1-076-21
Record Dates: First submitted 2021-10-08; First posted 2021-10-25 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Lumbar Facet Arthrosis; Nerve Degeneration
MeSH Terms: conditions — Nerve Degeneration | interventions — Shadowing Technique, Histology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The excess tissue harvested from the participants will be stored in the biorepository
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active group: Patients who are scheduled to undergo lumbar spinal surgery and fulfill the inclusion and exclusion criteria
  Interventions: Procedure: Spinal surgery; Other: Histology

INTERVENTIONS:
Procedure: Spinal surgery — In participants who undergo elective lumbar spinal surgery and consented for research, the medial branch and dorsal rami will be harvested for histological analysis.
Other: Histology — The harvested nerves will be fixed, cut into smaller sections. Analysis of macroscopic and light microscopic sections will be carried out

SUMMARY:
The purpose of the study is to understand the composition of the nerves supplying the facet joints in low back.

DETAILED DESCRIPTION:
After written informed consent, the nerves supplying the facet joints - lumbar dorsal rami and its medial branches, will be harvested when they are exposed during spinal surgery. These nerves will be fixed, washed and further dissected to enable smaller sections. The cut section will be stained and subjected to analysis of overall cross-sectional area and presence of connective tissue sheaths under light microscope.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18 or over
* be able to give informed consent
* scheduled to undergo lumbar spinal surgery

Exclusion Criteria:

* Children under 18 years old
* Vulnerable adults
* Adults with incapacity
* Inability to provide informed consent
* History of previous spinal surgery
* history of previous RF ablation for low back pain
* has COVID-19 or displaying symptoms of COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be the cohort of patients who are scheduled to undergo lumbar spinal surgery. The potential population will be identified from the patients who are being invited for the surgery. All prospective participants will be sent an invitation letter and Participant Information Sheet along with their the clinical appointment letters.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Nerve Histology | one year
  Percentage of nerves containing more than 50% sensory fibres in lumbar dorsal rami/medial branches to assess whether they are sensory or motor nerves

CONTACTS AND LOCATIONS:
Overall Officials: Saravanakumar Kanakarajan, MD FRCA, Principal Investigator — NHS Grampian
Locations (1):
- Woodend Hospital, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No